CLINICAL TRIAL: NCT03672682
Title: SMOLY : Phenotype and Functions of Monocyte Subtypes in High Grade B Lymphoma: Towards New Biomarkers?
Acronym: SMOLY
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_9799_SMOLY; 16.40 (Other: Comité d'Ethique Régional); 2043484 (Other: CNIL)
Record Dates: First submitted 2017-10-10; First posted 2018-09-14 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: DLBCL
Keywords: DLBCL; chemosensitivity; chemoresistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Patient selection from the BMS_LyTrans database
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DLBCL with chemoresistance: 15 patients with DLBCL with chemoresistance or relapsed less than 2 years after completion of first-line therapy
- DLBCL with chemosensitivity: 15 patients with DLBCL with chemosensitivity without relapse within 2 years following the end of first-line therapy.
- Healthy patients: 15 healthy patients

SUMMARY:
Large-cell B-cell lymphoma (DLBCL) is the most common non-Hodgkin's lymphoma and accounts for about 40% of new cases. Although the DLBCL is a single entity in the WHO classification, several subgroups with different prognoses are recognized. These subgroups take into account the tumor localization (primitive cerebral lymphoma, serous lymphoma, intravascular or exclusive lymph node) or a particular molecular signature (GCB profile, germline center B cell or ABC, activated B cell). Despite the introduction of immunotherapy, treatment failures are common. Overall survival at 5 years is estimated to be between 26 and 73%. This highlights the important heterogeneity of this pathology and therefore the need for biomarkers prognosis. Recently, an increase in monocytes in the blood of DLBCL patients has been proposed as a prognostic factor for independent survival. This marker of poor prognosis is also found in many solid.

Monocytes are effectors of the inflammatory response. They have different functional profiles depending on the level of expression of CD14 and CD16. Four subtypes of monocytes are distinguished: classical (CD14posCD16neg), intermediate (CD14posCD16pos) and non-classical (CD14lowCD16pos); the latter population is divided into two sub-groups depending on the expression of the SLAN protein. The different monocytic subpopulations have very diverse functions ranging from an immunosuppressive profile to an activation of the immune system. CD14posCD16neg monocytes are specialized in phagocytosis, production of oxygen derivatives (ROS) and pro-inflammatory cytokine secretion in response to microbial infection. CD14dimCD16pos monocytes are specialized in immune surveillance and produce proinflammatory cytokines such as TNFα and IL-1β in response to LPS stimulation.7 The Slanpos subpopulation produces IL-12 and thus has pro-inflammatory properties. Finally, CD14posCD16pos monocytes have controversial functions. For some authors, they produce the immunomodulatory cytokine IL-10, inhibit the proliferation of CD4 T lymphocytes and induce the recruitment of regulatory T lymphocytes, while for others they produce TNF-α, a pro- inflammatory.From a practical point of view CD14 and CD16 expression forms a continuum, which translates into complexity in the phenotypic definition of these cells and explains the contradictory data on their functionalities. Interestingly, in a laboratory work and in the course of publication, this fraction is increased in the blood of DLBCL patients compared to healthy donors (manuscript in preparation), on the contrary the monocytic fraction CD14dimCD16 pos is decreased in these patients.

In the end, if the increase in monocytes is known to be poor prognosis in patients with DLBCL, the monocyte fraction involved and the monocytic functions involved in this phenomenon are not known.

Since 2011, the Clinical and Biological Hematology Services have a database from a research protocol (BMS_LyTrans). This protocol includes patients with DLBCL as well as healthy patients, in order to allow the biological characterization of biomarkers in this pathology. Thus, we have blood samples and analysis of certain monocyte subtypes by flow cytometry at diagnosis, in more than 100 patients with DLBCL.

DETAILED DESCRIPTION:
Primary objective :

Describe and compare the distribution of the different monocytic subpopulations according to the chemosensitivity profile (group 1) or chemoresistance (group 2) of patients with DLBCL and healthy donors (group 3), and identify their specific functionalities.

Secondary objective :

To determine the prognostic impact in terms of progression-free survival (EFS) of the distribution of the monocytic sub-population (s) defined i during the primary objective, in a retrospective study (BMS Ly Trans)

Design/Methodology : Retrospective, observational, monocentric study.

1. - Part 1: Phenotypic and functional study of monocytic sub - populations of patients with DLBCL.

   - Patient selection from the BMS_LyTrans database : Group 1: 15 patients with DLBCL with chemoresistance or relapse less than 2 years after completion of first-line therapy.

   Group 2: 15 patients with DLBCL with chemosensitivity without relapse within 2 years following the end of first-line treatment.

   Group 3: 15 healthy patients.

   A - Irish Lab (Nashville)

   - Phenotypic analysis by mass cytometry: This new technology allows the integration of multiple data with membrane markers, intracytoplasmic proteins as well as transcription factors, thus providing global modeling of signaling pathways

   B - UMR 917 (Rennes) 8 months Cell sorting: The four subtypes of monocytes described above will be sorted by flow cytometry according to the expression of CD14, CD16 and Slan.

   - High-throughput transcriptional analysis: cell lysis and real-time PCR in order to study the expression of genes involved in the mechanisms of immunomodulation.Bio-informatics, Integrated analysis: The set of clinical, transcriptomic and proteomic data will be analyzed in an integrated way using tools and algorithms working within the Irish lab.
2. - 2nd part (Rennes) - 6 months : Populations differentially expressed between groups in part 1 will be analyzed on a cohort of 100 samples. These parameters will be analyzed jointly after integration in a database, uni- and multivariate analysis and the survival probability will be calculated for groups with a log-rank test.

Expected benefits :

1. - To allow a better understanding of the monocyte compartment in DLBCL, particularly with regard to the immunosuppressive capacity of some of these cellular subtypes.
2. - To refine the interest of the biomarker "monocyte level" on EFS in patients with DLBCL, highlighting the monocyte subtype involved.
3. - To continue the collaboration between the two sites, which will allow to combine technologies and expertise present in Rennes (patient recruitment, cell sorting, molecular analysis (Biomark)) or in Nashville (CyTOF, bioinformatics, integrated analysis).

ELIGIBILITY:
Inclusion Criteria:

* Age> or equal to 18 years and <or equal to 70 years
* Large cell diffuse NHL B (WHO)
* Stage I - II bulky with tumor mass> 7cm or stage III or IV of the Ann Arbor classification
* No prior treatment (even corticosteroid therapy)
* HIV negative
* Informed consent signed
* Patient follow-up> 2 years after completion of first-line treatment

Exclusion Criteria:

* Age <18 years or> 70 years
* Aggressive transformation of a known low-grade NHL
* Primary CNS Lymphoma
* MALT transformed lymphoma or Burkitt's lymphoma
* Lymphoma post transplantation
* Stage I or II with tumor mass <or equal to 7cm
* Cancer with the exception of carcinoma in situ of the cervix or non-invasive cutaneous epithelium
* History of cured cancer treated systematically and / or causing secondary complications in the six months prior to inclusion in the protocol
* Pre-treatment
* HIV positive
* Patient with a disability who does not have a good understanding of informed consent
* Unsigned informed consent
* Patient follow-up <2 years after completion of first-line treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient selection from the BMS_LyTrans database :
  Group 1: 15 patients with DLBCL with chemoresistance or relapse less than 2 years after completion of first-line therapy.
  Group 2: 15 patients with DLBCL with chemosensitivity without relapse within 2 years following the end of first-line treatment.
  Group 3: 15 healthy patients.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Proportion of monocytic sub-population(s) | At inclusion
  Increased proportion of one or more monocytic sub-populations (s) and / or modulation of the markers tested in one of the three groups studied.

SECONDARY OUTCOMES:
Progression-free survival | 2 years post diagnosis
  Difference of EFS in the validation cohort between patients with DLBCL having an increased proportion of one or more monocytic subpopulation (s) or modulation of the markers suspected in the descriptive phase, and the others.

CONTACTS AND LOCATIONS:
Locations (1):
- Rennes Univeristy Hospital, Rennes, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No